CLINICAL TRIAL: NCT02290236
Title: Monitored Saturation Post-ICU; Correlation to Charted Saturation, Pre-intensive Care Unit Obstructive Sleep Apnea and Outcome
Brief Title: Monitored Saturation Post-ICU
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, MD, PhD, Karolinska University Hospital
Other Study IDs: Post ICU Sat
Record Dates: First submitted 2014-10-06; First posted 2014-11-14 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Sleep Apnea, Obstructive; Respiratory Insufficiency
MeSH Terms: conditions — Sleep Apnea, Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulseoximetry — Peripheral saturation will be recorded continuously
  Other Names: Saturation

SUMMARY:
The overall aim with this project is to describe the correlation between measured and charted saturation after intensive care and also describe the saturation-pattern in these patients. The investigators will also correlate post-ICU desaturations measured as oxygen denaturation index and complications to pre-ICU obstructive sleep apnea and the STOP BANG screening questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.
* Admitted to the Central Intensive Care Unit (CIVA)
* Signed informed conscent by the patient or a relative

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are discharged from the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Oxygen desaturation index (ODI) | Days
  Measured by continuous pulseoximetry

SECONDARY OUTCOMES:
STOP Bang screening questionnaire | Days
  At inclusion the STOP BANG screening questionnaire will be completed

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Department of Anesthesiology, Surgical Services and Intensive Care Medicine, Karolinska University Hospital, Solna, Stockholm, Sweden